CLINICAL TRIAL: NCT02558452
Title: European Transplant Registry of Senior Renal Transplant Recipients Receiving Initial Immunosuppression With Tacrolimus Once Daily, Mycophenolate and Steroids
Brief Title: European Transplant Registry of Senior Renal Transplant Recipients on Advagraf
Acronym: SENIOR
Status: Not yet recruiting | Type: Observational
Sponsor: Klemens Budde (Other)
Collaborators: Dr. med. univ. L. J. Lehner (Unknown); Charite University, Berlin, Germany (Other); ERA-EDTA (Unknown); DESCARTES Working Group On Transplantation (Other); European Kidney Transplant Association (EKITA) (Other)
Responsible Party: Sponsor-Investigator, Klemens Budde, Prof. Dr. Klemens Budde, Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Other Study IDs: SENIOR
Record Dates: First submitted 2015-09-19; First posted 2015-09-24 (Estimated); Last update posted 2016-08-12 (Estimated); Status verified 2016-08

CONDITIONS: Graft Failure; Death; Acute Rejection of Renal Transplant; Infections; Bone Disease; Post Transplant Diabetes Mellitus; Quality of Life; HLA Antibody Production; Cardiovascular Risk Factors; Non-HLA Antibody Production
Keywords: elderly kidney transplant recipient; registry; tacrolimus once daily
MeSH Terms: conditions — Death; Infections; Bone Diseases | interventions — Mycophenolic Acid; Steroids

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples Without DNA — HLA antibodies, Non HLA antibodies
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Tacrolimus once daily (Advagraf) — Antibody induction by antithymocyte Globulin (ATG) or Basiliximab possible but not mandatory
  Other Names: mycophenolate; steroids

SUMMARY:
SENIOR transplant Registry European transplant registry of senior renal transplant recipients (above the age of 65 years) receiving initial immunosuppression with tacrolimus once daily, mycophenolate and steroids to investigate long term outcomes on an observational basis.

DETAILED DESCRIPTION:
The purpose of the registry is to establish data on the long-term outcome of elderly renal transplant recipients receiving an initial standard immunosuppression with tacrolimus once daily, mycophenolate and steroids The objectives of this registry are to investigate the long-term course of renal transplantation in the elderly European population (≥65 years) under immunosuppression with tacrolimus once daily, mycophenolate and steroids in order to better define risk factors for patient death and graft loss and predictors for favourable outcomes in this growing population.

For this purpose, the SENIOR transplant registry will be implemented to collect data on graft loss, death, renal function, quality of life and biopsy proven acute rejections (BPAR), analyze common complications such as severe infections, opportunistic infections (CMV and/or BKV viremia), malignancies, cardiovascular events, and hospitalisations in a large population of European senior renal allograft recipients. In addition, type and severity of rejections (Banff-grade, steroid resistant rejections, antibody-mediated rejections, antibody-treated rejections, recurrent rejections), development of circulating donor specific antibodies (DSA), cardiovascular risk factors (such as diabetes, development of posttransplant diabetes (PTDM), hypertension), renal function (as estimated by CKD-EPI), and proteinuria will be longitudinally assessed in parallel to immunosuppressive doses and drug levels. The registry will focus on common side effects of immunosuppressive therapy (such as leucopenia, anemia), treatment patterns and reasons for treatment changes. Finally, a prospective analysis of quality of life including the burden of medication in elderly transplant recipients is planned.

All recipients (≥65 years) of a kidney transplant who are willing to participate in the European SENIOR-Registry may enter the registry prior to transplantation if they are fulfilling all in- and none of the exclusion criteria and receive the intended initial immunosuppression consisting of tacrolimus once daily (Advagraf, initially adjusted to trough blood levels of ≥5ng/ml), mycophenolate (either ≥1.0g/day Mycophenolate Mofetil (MMF) or ≥720mg/d enteric-coated Mycophenolate Sodium (EC-MPS)) and Steroids.

There will be 12 study visits during the 10 year period. Except for quality of life questionnaires there are no study specific procedures planned. Only data will be recorded which anyway will be recorded in clinical routine.

The study population will consist of a representative group of approximately 1000 senior (≥65 years) kidney transplant patients, who receive a renal allograft and an initial standard triple immunosuppression (tacrolimus once daily (Advagraf), mycophenolate (either ≥1.0g/day Mycophenolate Mofetil (MMF) or ≥720mg/d enteric-coated Mycophenolate Sodium (EC-MPS)) and steroids. The patients will be recruited from approximately 42 transplant centers in Europe.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, aged ≥65 years
* Patients who received a renal allograft
* Patients who are willing and able to participate in the study and from whom written informed consent has been obtained
* Patients on an intended standard triple therapy with tacrolimus once daily (Advagraf with trough level ≥5ng/ml) in combination with mycophenolate (either ≥1.0g/day MMF or ≥720mg/d EC-MPS) and Steroids (≥5mg prednisolone or equivalent)
* Patient must have received primary or secondary renal allograft from a blood group compatible donor (either deceased or living)
* Patients with low to standard immunological risk, who had a PRA 20% (PRA testing according to center's practice) or no known donor specific antibodies at transplantation

Exclusion Criteria:

* Multi-organ recipients (solid organ or bone marrow)
* More than secondary renal allograft recipients
* Blood group A,B,O-incompatible allografts
* Documented presence of donor specific antibodies (DSA)
* Panel reactive antibody (PRA) >20% prior to transplantation (PRA testing according to center's practice)
* Patients having received any other induction therapy than Basiliximab or depleting polyclonal antithymocyte antibodies (ATG) (e.g. OKT3, Campath)
* Patients receiving Sirolimus, Everolimus, Azathioprine, Belatacept or Cyclophosphamide within 3 months prior to or at enrolment
* History of alcohol or drug abuse with less than 6 months of sobriety
* Patient with any condition that may affect absorption of immunosuppressives, (e.g. severe diarrhoea, gastrectomy, active peptic ulcer disease or clinically significant diabetic gastroenteropathy) or tacrolimus metabolism (e.g. liver cirrhosis)
* Patient with mental dysfunction or inability to cooperate within the study
* Patients who have been institutionalized by official or court order

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study population will consist of a representative group of approximately 1000 senior (≥65 years) kidney transplant patients, who receive a renal allograft and an initial standard triple immunosuppression (tacrolimus once daily (Advagraf), mycophenolate (either ≥1.0g/day Mycophenolate Mofetil (MMF) or ≥720mg/d enteric-coated Mycophenolate Sodium (EC-MPS)) and steroids. The patients will be recruited from approximately 42 transplant centers in Europe.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-12; Primary Completion 2027-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Patient survival | From date of transplantation until the date of death from any cause, assessed up to 10 years
Renal graft survival | From date of transplantation until the date of documented graft failure (need for permanent dialysis, explantation of the graft, retransplantation) or date of death from any cause, whichever came first, assessed up to 10 years
Biopsy proven acute rejection (BPAR) | Time of transplantation to date of first BPAR and consecutive BPARs, assessed up to 10 years
  Type of rejection according to BANFF 2013 classification
Development of anti-HLA antibodies | Time of transplantation to date of first detection of any HLA antibodies, assesments are month 3 and year 1,3,5,7 and 10 in the central laboratory and all in all up to 10 years locally
  type of antibodies (by HLA class and specificity), outcome after antibody production
Renal graft function by estimated glomerular Filtration rate (eGFR) by CKD-EPI) calculation | Assesment of renal graft function over time up to 10 years or graft failure or death, whichever comes first
  Change of creatinine from baseline to the discrete observational visits, Calculation of eGFR (CKD-EPI) and eGFR slope
Development of non-HLA antibodies | Time of transplantation to date of first detection of any HLA antibodies, assesments are month 3 and year 1,3,5,7 and 10 in the central laboratory and all in all up to 10 years locally
  type of antibodies, outcome after antibody production
Development of donor specific antibodies (DSA) | Time of transplantation to date of first detection of any HLA antibodies, assesments are month 3 and year 1,3,5,7 and 10 in the central laboratory and all in all up to 10 years locally
  type of antibodies (by HLA class and specificity), outcome after antibody production

SECONDARY OUTCOMES:
Incidence of kidney biopsies and suspected rejections | from time of transplantation for up to 10 years
  Incidence (number) of kidney biopsies and suspected rejections
Stroke | from time of transplantation up to 10 years
  number and type of events
Coronary revascularization procedure | from time of transplantation up to 10 years
  number and type of events
Carotid surgery | from time of transplantation up to 10 years
  number and type of events
Revascularisation procedures for symptomatic peripheral artery disease | from time of transplantation up to 10 years
  number and type of events
Symptomatic peripheral artery disease | from time of transplantation up to 10 years
  number and type of Events, classification by Fontaine
cardiac death | from time of transplantation to the date of the event for up to 10 years, whichever comes first
  number and type of events
non-fatal myocardial infarction | from time of transplantation to the date of the event for up to 10 years, whichever comes first
  number and type of events
Hospitalisations | from time of transplantation up to 10 years
  Incidence of hospitalisations, reasons and length of hospitalisations
Infections in general | from time of transplantation up to 10 years
  Incidence of infections and type of infections
Cytomegalovirus (CMV) disease | from time of transplantation up to 10 years
  Incidence, defined by symptomatic CMV infection (including pulmonary and intestinal infections)
CMV infection | from time of transplantation up to 10 years
  Incidence, Defined by nucleic acid testing (NAT) in blood
BKV (BK-Virus) infection | from time of transplantation up to 10 years
  Incidence; Def: NAT testing in urine and blood or by biopsy staining
Pneumocystis jiroveci pneumonia infection | from time of transplantation up to 10 years
  Incidence
Malignancies | from time of transplantation up to 10 years
  Incidence, types of malignancies
Post transplant diabetes mellitus | from time of transplantation up to 10 years
  Incidence and time to development of posttransplant diabetes mellitus (PTDM)
Immunosuppressants | from time of transplantation up to 10 years
  Type of IS, Changes of IS
Bone disease | from time of transplantation up to 10 years
  number of fractures, measured height (meters)
Quality of life measures | from time of transplantation up to 10 years
  Quality of life by questionnaire (SF36, MTSODS)

CONTACTS AND LOCATIONS:
Overall Officials: Lukas J Lehner, MD, Principal Investigator — Charite University, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
aggregated data are available through the Steering committee of DESCARTES and EKITA